CLINICAL TRIAL: NCT02881918
Title: Anti-tumor Specific Immune Response in Head and Neck Cancers
Acronym: CORISAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2016 / CORISAT-GALLET/SR
Record Dates: First submitted 2016-08-19; First posted 2016-08-29 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- squamous cell carcinoma: Patients affected by Head & Neck Squamous Cell Carcinoma. Blood sample at diagnosis, before any antitumor treatment
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood sample with 6 tube of blood (40 mL), after diagnosis and before any specific anticancer treatment

SUMMARY:
The purpose is the description of anti-tumor immune responses in general and according to clinical stage and disease free survival (DFS: survival without recurrence (local or distant)) in patients with Head & Neck Squamous Cell Carcinoma

Secondary purposes are:

* Study of relationship between anti-tumor immune response and qualitative (yes/no) and quantitative (number) presence of circulating tumor cells (CTCs);
* Study of relationship between qualitative (yes/no) and quantitative (number) presence of CTCs and clinical stage as well as DFS
* Study of relationship between anti-tumor immune response and clinical stage as well as DFS.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Head & Neck Squamous Cell Carcinoma after extension assessment, regardless of clinical stage (TNM UICC stage I-IV), before any medical or surgical treatment specifically directed against cancer (radiotherapy, surgery, chemotherapy or targeted therapy)
* Consent to participate to the study, non-opposition
* Affiliation to social security

Exclusion Criteria:

* History of neoplasia, synchronous cancer, auto-immune disease, organ transplantation, chemotherapy
* HIV infection
* Corticotherapy during 15 days before blood sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Head & Neck Squamous Cell Carcinoma before any medical or surgical treatment specifically directed against cancer
Sampling Method: Non-Probability Sample
Enrollment: 154 (Estimated)
Dates: Start 2017-03-14 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of spontaneous responses against tumor-associated antigens (TAA) according to tumor stage | day 0

SECONDARY OUTCOMES:
Functional signature of T cell responses (polyfunctionality index of lymphocytes) according to tumor stage | day 0
  Effector functions and phenotypes of T cells
Number of CTCs according to tumor stage | day 0
Polyfunctionality index of lymphocytes according to number of CTCs | day 0
Disease free survival (survival without local or distant recurrence) according to Presence pr absence of CTCs at diagnosis | 2 years after diagnosis
Disease free survival (survival without local or distant recurrence) according to Presence or absence of spontaneous responses against TAA | 2 years after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Patrice GALLET, Principal Investigator — Service de ORL, Institut Louis Mathieu, CHRU de Nancy
Locations (6):
- France (6):
  - Service d'ORL - CHRU BESANCON, Besançon
  - Service d'ORL - CHRU DIJON, Dijon
  - Service d'ORL - CHRU REIMS, Reims
  - Service d'ORL - CHRU STRASBOURG, Strasbourg
  - Institut de Cancérologie Alexis Vautrin, Vandœuvre-lès-Nancy
  - Service ORL - Institut Louis Mathieu - CHRU NANCY, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No